CLINICAL TRIAL: NCT01743287
Title: A Six-month, Multi Center, Randomized, Double Blind, Parallel-group, Placebo Controlled Study to Evaluate Efficacy and Safety of Imotun Capsule in Osteoarthritis of the Knee
Brief Title: The Study to Evaluate Efficacy and Safety of Imotun Capsule in Osteoarthritis of the Knee
Acronym: ABSOLUTE-OS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 238KOA12F
Record Dates: First submitted 2012-12-03; First posted 2012-12-06 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis of the knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imotun capsule (Experimental): Imotun capsule: 300.03mg/cap, orally, 1 capsule once a day during 24 weeks
  Interventions: Drug: Imotun capsule
- Imotun capsule placebo (Placebo Comparator): Imotun capsule Placebo: Placebo 1 capsule once a day during 24 weeks
  Interventions: Drug: Imotun capsule placebo

INTERVENTIONS:
Drug: Imotun capsule — Imotun capsule: Avocado-Soya Unsaponifiables 300.03mg/Cap, per oral, a capsule once a day during for 24 weeks
  Arms: Imotun capsule
Drug: Imotun capsule placebo — Imotun capsule placebo: per oral, a capsule a day during 24 weeks
  Arms: Imotun capsule placebo

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of Imotun capsule in osteoarthritis of the knee

DETAILED DESCRIPTION:
This is a six-month, multicenter, randomized, double blind, parallel-group,placebo controlled study. Patients take Imotun capsules or placebo once a day, between the meals. Patients are allowed to take study drugs during the meal in the case of intolerant reflux of oil smell from GI. If patients do not tolerate the pain, they are able to take Celecoxib as a rescue medication during 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients who aged 40 or more and agreement with written informed consent
* Patients with osteoarthritis according to ACR criteria lasted for the past 3 months or more
* Patients with Kellgren & Lawrence grade Ⅱ~Ⅲ on radiographs
* Patients with 40mm or higher 100mm Pain VAS on screening and baseline visit (based on more painful knee)
* Patients with Lequesne's index 5 or more on screening and baseline visit

Exclusion Criteria:

* Patients who had taken SYSADOA within the past 3 months (Imotun, diacerein, s-adenosyl-methionone, JOINS, glucosamine, chondroitin and any other cartilage protective agents determined by investigator)
* Patients who experienced cartilage surgery within the past 5 years or arthroscope surgery within a year(one side or both)
* Patients who were treated with joint space injection within the past 3 months
* Patients who had taken NSAIDs including pain killers within 7 days (except, it is acceptable to enroll the study if the patients have wash out periods at least 7 days before randomization)
* Patients with hypersensitivity or allergy to the study or rescue medicine or those who have medical history.
* Patients with severe liver, kidney or cardiac diseases who are not acceptable for the study determined by investigator
* Patients with active peptic ulcer or GI bleeding.
* Pregnancy, nursing women or women of reproductive age who do not agree to the contraception.
* Patients with abuse of alcohol, illegal drugs or drug dependency
* Patients who were treated with another investigational product within the past 4 weeks
* All other patients who are not acceptable for the study determined by investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2012-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
100mm pain VAS | 24 weeks
  assessment of the 100mm pain VAS
change from baseline Lequesne's index score at 24 weeks | baseline, 24 weeks

SECONDARY OUTCOMES:
change from baseline Lequesne's index score at 4 weeks | baseline, 4 weeks
change from baseline 100mm pain VAS at 4 weeks | baseline, 4 weeks
100mm pain VAS | 4 weeks
  assessment of 100mm pain VAS
global assessment | 4 weeks
  global assessment by physician and patient
administration days of the rescue medication | 24 weeks
The rate of patients who consumed the rescue medication | 24 weeks
change from baseline Lequesne's index score at 8 weeks | baseline, 8 weeks
change from baseline Lequesne's index score at 16 weeks | baseline, 16 weeks
change from baseline 100mm pain VAS at 8 weeks | baseline, 8 weeks
change from baseline 100mm pain VAS at 16 weeks | baseline, 16 weeks
change from baseline 100mm pain VAS at 24 weeks | baseline, 24 weeks
100mm pain VAS | 8 weeks
  assessment of 100mm pain VAS
100mm pain VAS | 16 weeks
  assessment of 100mm pain VAS
global assessment | 8 weeks
  global assessment by physician and patient
global assessment | 16 weeks
  global assessment by physician and patient
global assessment | 24 weeks
  global assessment by physician and patient
dosing quantity of the rescue medication | 24 weeks

OTHER OUTCOMES:
rate of adverse event | up to 24 weeks
laboratory test | up to 24 weeks
medication history | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Myung Chul Lee, phD, Principal Investigator — Seoul National University Hospital
Locations (10):
- South Korea (10):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheonbuk-do
  - Inje University Busan Paik Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Chonnam National University Hwasun hospital, Hwasun
  - Chonbuk National University Hospital, Jeonju
  - Bundang CHA medical center, Seongnam
  - Seoul National University Hospital, Seoul
  - KyungHee University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - ASAN Medical Center, Seoul